CLINICAL TRIAL: NCT01583842
Title: 124I-Metaiodobenzylguanidine (MIBG) PET/CT Diagnostic Imaging and Dosimetry for Patients With Neuroblastoma: A Pilot Study
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Funding
Sponsor: Miguel Pampaloni (Other)
Collaborators: Molecular Insight Pharmaceuticals, Inc. (Industry); Jubilant DraxImage Inc. (Industry)
Responsible Party: Sponsor-Investigator, Miguel Pampaloni, Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 12088; NCI-2012-00617 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2012-04-17; First posted 2012-04-24 (Estimated); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Neuroblastoma
Keywords: neuroblastoma; imaging; 124I-MIBG; 131I-MIBG; PET/CT
MeSH Terms: conditions — Neuroblastoma | interventions — 3-Iodobenzylguanidine; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 124I-MIBG no-carrier added (Experimental): Patients are 3 years of age and older with relapsed or refractory neuroblastoma who are currently enrolled on a treatment protocol with 131I-MIBG.
  Interventions: Drug: 124I-Metaiodobenzylguanidine (MIBG) (no-carrier added); Procedure: Positron Emission Tomography (PET) /Computerized tomography (CT)
- 124I-MIBG carrier added (Experimental): Patients are 3 years of age and older with relapsed or refractory neuroblastoma who are currently enrolled on a treatment protocol with 131I-MIBG.
  Interventions: Drug: 124I-MIBG (carrier added); Procedure: Positron Emission Tomography (PET) /Computerized tomography (CT)
- Imaging Only (Active Comparator): Participants with high-risk neuroblastoma will receive imaging only without 124I-MIBG
  Interventions: Procedure: Positron Emission Tomography (PET) /Computerized tomography (CT)

INTERVENTIONS:
Drug: 124I-Metaiodobenzylguanidine (MIBG) (no-carrier added) — 124I-MIBG (no-carrier added) Administration (infusion, 1-2 minutes) followed by sequential PET/CT dosimetry scans on Days 0, 1, 2 and 5.
  Optional 124I-MIBG (no-carrier added) Administration & PET/CT scan 6 weeks later.
  Other Names: 124I MIBG; MIBG
  Arms: 124I-MIBG no-carrier added
Drug: 124I-MIBG (carrier added) — 124I-MIBG (carrier added) Administration (infusion, 60 minutes) followed by sequential PET/CT dosimetry scans on Days 0, 1, 2 and 5.
  Optional 124I-MIBG (carrier added) Administration & PET/CT scan 6 weeks later.
  Other Names: 124I MIBG; MIBG
  Arms: 124I-MIBG carrier added
Procedure: Positron Emission Tomography (PET) /Computerized tomography (CT) — A PET scan measures important body functions, such as metabolism. CT imaging uses special x-ray equipment, and in some cases a contrast material, to produce multiple images of the inside of the body. Combined PET/CT scans combine the processes of both a PET and CT at the same time.
  Other Names: PET/CT

SUMMARY:
This is a pilot study with the primary purpose to describe organ dosimetry and acute toxicities using no carrier added and carrier added 124I-MIBG PET/CT in patients with neuroblastoma (NB). Eligible patients are 3 years of age and older with relapsed or refractory neuroblastoma who are currently enrolled on a treatment protocol with 131I-MIBG. After all eligibility criteria are met, patients will receive a diagnostic imaging dose of 124I-MIBG followed by sequential PET/CT dosimetry scans on Days 0, 1, 2 and 5. Subsequent, planned therapeutic administration of 131I-MIBG will occur between Days 7 to 21, as specified by the patient's therapeutic MIBG protocol. An optional single follow up 124I-MIBG PET-CT scan will be done to assess tumor sites 6 weeks after the patient has their MIBG therapy.

DETAILED DESCRIPTION:
Accurate radiation dose evaluation is important in patients with malignant tumors, and this is especially critical in children with NB who will be receiving several dose of therapeutic 131I. The accurate quantification of the isotope-labeled analog can only be achieved by using positron emission compounds, such as 124I. Unlike planar images, which were used to obtain kinetic information, and SPECT reconstruction modalities that were aimed to assess the spatial distribution of radioactivity, 3D PET imaging-based dosimetry is a method which provides a more accurate estimation of the cumulated radioactivity distribution. Because PET provides better quantitative accuracy, when compared to SPECT regarding the tissue absorbed information, we hypothesize PET would better correspond with tumor response and normal organ toxicity. Early studies using I-124 for dosimetry in thyroid cancer have been promising.

Demonstration of the feasibility and accuracy of this new imaging modality, with the excellent prospect for more accurate dosimetry, will improve tumor localization and optimize therapeutic dosing with 131I-MIBG. The results of our work may potentially have also implications in the study of other neuroendocrine tumors. The Section of Nuclear Medicine and the Laboratory of Functional Imaging at the University of California, San Francisco, are equipped with state of the art instruments and is run by a highly skilled staff which will guarantee the success of the proposed research.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be >/= 3 years of age and able to cooperate for the PET CT scan when registered on study.
* Patients must have a diagnosis of neuroblastoma either by histologic verification of neuroblastoma and/or demonstration of tumor cells in the bone marrow with increased urinary catecholamine metabolites.
* Recurrent/progressive disease at any time. Biopsy is not required, even if there is a partial response to intervening therapy or
* Refractory disease (i.e. less than a partial response to frontline therapy, including a minimum of 4 cycles of chemotherapy). No biopsy is required for eligibility for this study.
* 123I-MIBG Uptake: Patients must have MIBG evaluable disease which is defined as evidence of uptake into tumor at one site within 4 weeks prior to entry on study and subsequent to any intervening therapy.
* Patients must meet eligibility criteria for 131I-MIBG therapy in order to participate in the dosimetry portion.
* All post-menarchal females must have a negative beta-Human Chorionic Gonadotropin (hCG) within 2 weeks prior to receiving the dose of 124I-MIBG. Males and females of childbearing potential must practice an effective method of birth control while participating on this study, to avoid possible damage to the fetus.

Imaging only cohort:

- Patients with high-risk neuroblastoma are eligible at any time (during initial treatment or during treatment of relapsed/refractory disease) as long as they meet the requirements.

Exclusion Criteria:

* Pregnancy or lactating with the intent of breast feeding.
* Patients who require general anesthesia for MIBG imaging studies.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-04-09 (Actual); Primary Completion 2021-02-25 (Actual); Study Completion 2021-02-25 (Actual)

PRIMARY OUTCOMES:
Measurements of organ dosimetry using high specific activity (no carrier added) | Up to 7 weeks
  Descriptive statistics for each organ dose obtained from the organ dosimetry data will be reported, to demonstrate organ dosimetry calculations are feasible and concordant with prior calculations in prior conjugate planar dosimetry imaging studies and our pre-clinical murine models
Measurements of organ dosimetry using low specific activity (carrier added) | Up to 7 weeks
  Descriptive statistics for each organ dose obtained from the organ dosimetry data will be reported, to demonstrate organ dosimetry calculations are feasible and concordant with prior calculations in prior conjugate planar dosimetry imaging studies and our pre-clinical murine models
Number of participants with grade 3 or 4 imaging-related toxicities. | Up to 7 weeks
  All patients will have toxicity monitoring for 6 weeks following 124I-MIBG administration. Toxicities will be graded according to the NCI Common Toxicity Criteria for Adverse Events (CTCAEv4.0)and attribution assigned.
Change from baseline of blood pressure | Up to 7 weeks
  Blood pressure will be recorded before, during, end injection and post-injection at baseline, days 1, 2 and 5 and again at week 7 if participants choose to have optional week 7 scan
Change from baseline of pulse measurements | Up to 7 weeks
  Participants pulse will be recorded before, during, end injection and post-injection at baseline, days 1, 2 and 5 and again at week 7 if participants choose to have optional week 7 scan

SECONDARY OUTCOMES:
Measurements of tumor dosimetry using low specific activity (carrier added) | Up to 7 weeks
  Descriptive statistics will be used to report the tumor dosimetry data
Measurements of tumor dosimetry using high specific activity (no carrier added) | Up to 7 weeks
  Descriptive statistics will be used to report the tumor dosimetry data
Assessment of the accuracy of tumor imaging | Up to 7 weeks
  Descriptive statistics will be used to report the tumor dosimetry data compared to using 123I-MIBG scan with 3-dimensional imaging by SPECT or SPECT/CT

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Matthay, MD, Principal Investigator — University of California, San Francisco; Jose Miguel Hernandez-Pampaloni, MD, PhD, Principal Investigator — University of California, San Francisco; Youngho Seo, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No